CLINICAL TRIAL: NCT06380426
Title: A Multicenter Pharmacoepidemiological Cohort on Real Life Use of WEGOVY (Semaglutide) in Obese Patients With Monogenic Obesity
Brief Title: Real-life Evaluation of WEGOVY (Semaglutide) Treatment in Adults With Monogenic Obesity (ObGeSema)
Acronym: ObGeSema
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230441; IDRCB : 2023-A02003-42 (Other: ANSM)
Record Dates: First submitted 2024-04-11; First posted 2024-04-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Monogenic Obesity
Keywords: Monogenic obesity; Semaglutide; WEGOVY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Rare genetic forms of obesity, so called monogenic obesity are linked to alteration in energy balance involving hypothalamic pathways.

More than 60 genes encoding for proteins located in the hypothalamic leptin/melanocortin pathway have been described in the French National Protocol for Diagnostic and Care (PNDS).

The natural history of monogenic obesity is characterized by an early onset in childhood, with a major increase in weight in adolescence and young adulthood. The worsening of obesity exposes these patients to severe complications.

Severe obesity and eating disorders have a major impact on the quality of life of the person but also of the family and caregivers. Clinical management is complex and requires comprehensive, specialized and multidisciplinary management. But the usual lifestyle approaches have so far shown disappointing results, similarly to bariatric surgery which leads to a more frequent weight regain in the situation of monogenic obesity, justifying new approaches.

In this context, evaluating the response to treatment in the particular condition of monogenic obesity is crucial to propose therapeutic options as early as possible to limit weight evolution and its complications.

GLP-1 (glucagon-like peptide 1) based innovative therapies have recently emerged as a promising option for treatment of obesity and its complications. This is the case for Semaglutide 2.4mg/week (WEGOVY®), developed by Novo Nordisk. However, there is a lack of data to confirm that semaglutide could be also effective in monogenic obesity.

The hypothesis in this study is that treatment with Semaglutide 2.4mg/week (WEGOVY®) could be as effective in monogenic obesities as in common obesity.

DETAILED DESCRIPTION:
Rare genetic forms of obesity, so called monogenic obesity are linked to alteration in energy balance involving hypothalamic pathways. More than 60 genes encoding for proteins located in the hypothalamic leptin/melanocortin pathway have been described in the French National Protocol for Diagnostic and Care (PNDS).

The natural history of monogenic obesity is characterized by an early onset in childhood, with a major increase in weight in adolescence and young adulthood. The worsening of obesity exposes these patients to severe complications. Severe obesity and eating disorders have a major impact on the quality of life of the person but also of the family and caregivers. Clinical management is complex and requires comprehensive, specialized and multidisciplinary management. But the usual lifestyle approaches have so far shown disappointing results, similarly to bariatric surgery which leads to a more frequent weight regain in the situation of monogenic obesity, justifying new approaches.

In this context, evaluating the response to treatment in the particular condition of monogenic obesity is crucial to propose therapeutic options as early as possible to limit weight evolution and its complications.

GLP-1 (glucagon-like peptide 1) based innovative therapies have recently emerged as a promising option for treatment of obesity and its complications. This is the case for Semaglutide 2.4mg/week (WEGOVY®), developed by Novo Nordisk. However, there is a lack of data to confirm that semaglutide could be also effective in monogenic obesity.

The hypothesis in this study is that treatment with Semaglutide 2.4mg/week (WEGOVY®) could be as effective in monogenic obesities as in common obesity.

This study is a multicenter study which involves French largest Specialized Obesity Centers (CSO) (among which the APHP coordinating center) All adult patients with a genetic diagnosis of obesity to whom Wegovy is proposed, as part of the WEGOVY® early access and/or commercialization, or for whom Wegovy has already been initiated will be proposed to participate to the study. This also includes any patient having initiated the treatment and already having interrupted it, for any reason.

After the information has been done, the patient or guardian gives to the physician their oral non-opposition for the study that is recorded in the medical records.

This study will take advantage of WEGOVY's pre-marketing, early access authorisation and/or commercialization in France to set up a longitudinal follow-up of patients with monogenic obesity receiving Semaglutide.

Patients already treated with semaglutide at the time of study start (i.e. patients having initiated the treatment in the Early Access programme) will be included and followed-up, whereas inclusion and prospective follow-up of newly treated patients will only begin when Semaglutide becomes officially available.

The aim of the ObGeSema project is to set up a cohort composed of patients (1) having already initiated a treatment and (2) newly treated by Semaglutide in 14 Specialized Obesity Centres (CSOs) and describe their evolution over a 4 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (≥18 years)having already initiated a treatment with SEMAGLUTIDE (WEGOVY®) or with a physician's decision to initiate treatment in the standard care in the near future. All patients having initiated a treatment will be proposed to participate, including those having already stopped the treatment at the time of study initiation.
* Confirmation of monogenic obesity, as practiced in clinical routine, by the presence of a pathogenic or likely pathogenic variant in a gene with leptin-melanocortin pathway described in PNDS (https://www.has-sante.fr/jcms/p_3280217/fr/generique-obesites-de-causes-rares)
* Patients duly informed and not objecting to participate in the study
* Patients affiliated to a social security scheme or State Medical Assistance (AME).

Exclusion Criteria:

* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with monogenic obesity due to a pathogenic variant already treated or with the physician's decision to initiate treatment with Semaglutide 2.4mg/week (WEGOVY®) in the standard care. Patients under legal protection and State Medical Assistance (AME) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in weight and Body Mass Index (BMI) | From baseline (T0) to T12
  Percentage of subjects with a change in weight and Body Mass Index (BMI).Weight will be measured at initiation and at 12 months of the Wegovy treatment

SECONDARY OUTCOMES:
Change in weight and Body Mass Index (BMI) | From baseline (T0) to 6 and/or 24 and/or 36 and/or 48 and/or 60 months
  Percentage of subjects with a change in weight and Body Mass Index (BMI). Weight will be measured at initiation of the Wegovy treatment and at each visit
Reduction of body weight equal to or above 5% | From baseline (T0) to 6 and/or 12 and/or 24 and/or 36 and/or 48 and/or 60 months
  Percentage of subjects achieving a reduction of body weight equal to or above 5%(number of subjects with a % of body weight changes > -5%)X100/ number of the total subject
Change in Hunger score | From baseline (T0) to 12 and/or 24 and/or 36 and/or 48 and/or 60 months
  Number and percentage of subjects with change in Hunger score
Change in eating behaviour measured by Food Craving questionnaire | From baseline (T0) to 12 months
  Number and percentage of subjects with change in Food Craving scale
Change in eating behaviour measured by the Binge Eating Scale (BES) | From baseline (T0) to 12 months
  Number and percentage of subjects with change in Binge Eating Scale (BES)
Change in eating behaviour measured by the Dutch Eating Behaviour Questionnaire (DEBQ) | From baseline (T0) to 12 months
  Number and percentage of subjects with change in Dutch Eating Behaviour Questionnaire (DEBQ)
Change in eating behaviour measured by the Dykens questionnaire | From baseline (T0) to 12 months
  Number and percentage of subjects with change in Hyperphagia score with the Dykens questionnaire for intellectual disability
Change in eating behaviour measured by the Child Eating Behaviour Questionnaire (CEBQ) | From baseline (T0) to 12 months
  Number and percentage of subjects with change in the Child Eating Behaviour Questionnaire (CEBQ) for intellectual disability
Change in the International physical activity questionnaire (IPAQ - short form) | From baseline (T0) to 12 months
  Number and percentage of subjects with change of the International physical activity
Change in Digestive disorders (GIQLI ) | From baseline (T0) to 12 and/or 24 and/or 36 and/or 48 and/or 60 months
  Number and percentage of subjects with change in Digestive disorders (GIQLI ). Digestive disorders are measured by the Gastrointestinal Quality of Life Index (GIQLI)
Change in sleep disorder (MCTQ score) | From baseline (T0) to 12 months
  Number and percentage of subjects with Change in sleep disorder. Sleep disorder is measured with the Micro Munich Chronotype Questionnaire (MCTQ)
Change in score of quality of life scores (patient and parents) | From baseline (T0) to 12 months
  Number and percentage of subjects with change in score of quality of life scores .Quality of life is measured with the Impact of Weight on Quality of Life-Lite scale (IWQOL-Lite)
Change in anxiety and depression score | From baseline (T0) to 12 and/or 24 and/or 36 and/or 48 and/or 60 months
  Number and percent of subjects with change in anxiety and depression score. Anxiety and depression is measured with the Hospital Anxiety and Depression scale (HAD)
Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | From baseline (T0) to 6 and/or 12 and/or 24 and/or 36 and/or 48 and/or 60 months
  Number of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Christine POITOU-BERNERT, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris; Béatrice DUBERN, MD,PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Centre de référence Syndrome de Prader-Willi et autres obésités avec troubles du comportement alimentaire (PRADORT). Service de Nutrition, GH Pitié-Salpêtrière, APHP, Paris
  - CHU Pitié Salpêtrière - APHP, Paris

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodological sound proposal.